CLINICAL TRIAL: NCT07015684
Title: Open-label, Single-Center, Phase 1 Study to Estimate the Minimum Effective Dose (MED) of 131I-apamistamab for Non-myeloablative Conditioning in Patients With Severe Sickle Cell Disease
Brief Title: 131I-apamistamab-based Conditioning for Hematopoietic Stem Cell Transplant (HSCT) in Advanced Sickle Cell Disease (SCD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Actinium Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Markus Mapara, Professor of Medicine, Director of Bone Marrow Transplantation & Cell Therapy Program, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV1172
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Sickling Disorder Due to Hemoglobin S
Keywords: severe sickle cell disease; severe SCD; sickle cell disease; sickle cell; advanced SCD; advanced sickle cell disease; anemia; sickle cell disorders; hemoglobin S (HbS) Disease; Hemoglobin S Disease
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia; Sickle Cell Trait; Disease | interventions — Iodine; Sirolimus; Alemtuzumab; Whole-Body Irradiation; Exchange Transfusion, Whole Blood

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 131I-apamistmab-based nonmyeloablative conditioning (Experimental): Ten days before participants receive donor stem cell infusion, they will receive a dose of 131 I-apamistamab as an intravenous (IV) infusion into a vein in the arm. The 131 I-apamistamab product will be formulated in advance of the anticipated infusion date, for infusion on a specific date, based on target dose (100 mCi or 150 mCi, based on dose level).
  Interventions: Drug: 131I-apamistmab; Drug: Sirolimus; Drug: Campath; Drug: Total Body Irradiation; Procedure: Exchange Transfusion; Radiation: Planar gamma imaging

INTERVENTIONS:
Drug: 131I-apamistmab — 131I-apamistamab is a drug construct consisting of the apamistamab monoclonal antibody (mAb) and radioactive isotope iodine 131 (131I). The study drug will be patient-specific and will be manufactured for dosing on a specific date. The antibody dose will be at least 0.5mg/kg, however the final antibody amount may be higher if necessary based on the target radioactivity level. The 131I-apamistamab study drug requires patient details such as height, weight, a calculation to determine weight for use in calculating antibody amount for the dose. 131I-apamistmab will be given via intravenous (IV) infusion.
  Other Names: Iodine (131I) apamistamab
Drug: Sirolimus — Sirolimus is a macrocyclic lactone produced by Streptomyces hygroscopicus. It is an immunosuppressant agent. Sirolimus is to be given orally either as tablet or solution form. Dosage will be adjusted to a therapeutic target of 10-15 ng/mL in first 6 months post-transplant and 5-10 ng/mL after 6 months.
  Other Names: Rapamycin; Rapamune
Drug: Campath — Campath is a recombinant DNA-derived humanized monoclonal antibody that is directed against the 21-28 kD cell surface glycoprotein, CD52. CD52 is expressed on the surface of normal and malignant B and T lymphocytes, NK cells, monocytes, macrophages, and tissues of the male reproductive system. Campath will be given via IV at a total dose of 1 mg per kilogram of body weight.
  Other Names: Alemtuzumab
Drug: Total Body Irradiation — Radiation dose is 3Gy (Gy is a radiation unit of measurement). Radiation source and dose rates will be according to institutional practice. Total Body Irradiation (TBI) may be delivered from either linear accelerator or Cobalt sources.
  Other Names: TBI
Procedure: Exchange Transfusion — Patient will undergo a red blood cell (RBC) exchange transfusion to achieve a Hemoglobin S (HgbS) level < 20% prior to starting therapy to prevent the development of a vaso-occlusive Crisis (VOC).
Radiation: Planar gamma imaging — Dosimetric imaging will be performed using quantitative planar gamma camera acquisition. Planar gamma imaging is a technique used in medical imaging to take pictures of the inside of the body, particularly to look at how certain organs or tissues are functioning. This allows the study doctor to evaluate how the study drugs are absorbed into the body.
  Other Names: therapeutic radiation

SUMMARY:
The purpose of this study is to find the smallest amount of the 131 I-apamistamab needed for preparing patients with severe sickle cell disease (SCD) for a bone marrow transplant. This is the first time 131 I-apamistamab is being used for advanced Sickle Cell Disease (SCD) in the setting of allogeneic stem cell transplant. 131 I-apamistamab is an investigational product. This means that 131 I-apamistamab has not been approved by the Food and Drug Administration (FDA) for medical use in patients.

The study treatment that is given before the transplant is called the conditioning regimen. In this study, the investigators are adding a drug called 131 I-apamistamab instead of the conditioning regimen typically given before a stem cell transplant.

DETAILED DESCRIPTION:
The purpose of this study is to research the minimum effective dose (MED) of 131 I-apamistamab conditioning for hematopoietic stem cell transplantation for patients with advanced SCD. 131 Iapamistamab is an investigational product. This means that 131 I-apamistamab has not been approved by the Food and Drug Administration (FDA) for medical use in patients.

The study treatment that is given before the transplant is called the conditioning regimen. In this study, investigators are adding 131 I-apamistamab instead of the conditioning regimen typically given before a stem cell transplant.

The current standard of care conditioning for allogeneic stem cell transplant in SCD is a combination of chemotherapy, total body irradiation and an antibody called Campath. This study is being done to see if the stem cell transplant for SCD can still be effective by eliminating total body irradiation from the conditioning as it has potential long term side effects such as secondary cancers, infertility, early cataracts and lung toxicity.

This is a single center, Phase I, dose finding study to estimate the MED of hematopoietic stem cell transplantation for patients with advanced sickle cell disease using 131I-apamistmab-based nonmyeloablative conditioning. The study will enroll 24 patients who are 12-50 years of age with sickle cell anemia (Hb SS, SC, or Sβ0 thalassemia) and have an available HLA-matched sibling donor.

ELIGIBILITY:
Inclusion Criteria:

* Availability of an HLA-matched sibling donor
* Patients with sickle cell anemia (Hb SS, Sβ0 thalassemia or severe SC) who are 12 - 50 years of age inclusive AND who have 1 or more of the following:

  1. Clinically significant neurologic event (stroke) or any neurological deficit lasting at least 24 hours. Stroke will be defined as a clinically significant neurologic event that is accompanied by an infarct on cerebral MRI or cerebral arteriopathy requiring chronic transfusion therapy.
  2. History of two or more episodes of ACS in the 2-year period preceding enrollment despite supportive care measures (i.e. asthma therapy and/or hydroxyurea).
  3. History of three or more severe vaso-occlusive pain crises per year in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. a pain management plan and/or treatment with hydroxyurea).
  4. Administration of regular RBC transfusion therapy, defined as receiving 8 or more transfusions per year for 1 year or more to prevent vaso-occlusive clinical complications (i.e. pain, stroke, and ACS)
  5. An echocardiographic finding of tricuspid valve regurgitant jet (TRJ) velocity > or equal to 2.7 m/sec or pulmonary hypertension diagnosed by right heart catherization.
  6. Sickle hepatopathy defined as EITHER ferritin >1000mcg/L OR direct bilirubin >0.4mg/dl but <5xULN AND platelet count <250,000/uL at baseline
* Adequate organ functions as defined as:

  1. ECOG performance status of 2 or better
  2. Cardiac function: LVEF of 40% or greater
  3. Pulmonary Function: Pulse oximetry with a baseline oxygen saturation of 85% or greater and corrected DLCO of 40% or greater
  4. Hepatic Function: Serum conjugated (direct) bilirubin less than 5x upper limit of normal for age as per local laboratory, ALT and AST less than 5 x upper limit of normal as per local laboratory. Patients whose hyperbilirubinemia is the result of hyperhaemolysis, or a sever drop in hemoglobin post blood transfusion are not excluded.
  5. Absence of liver cirrhosis, bridging fibrosis and active hepatitis as documented by liver biopsy for patients with evidence of iron overload by serum ferritin or MRI. The histological grading and scale described by Ishak and colleagues (1995) will be used.

Donor Eligibility and Selection Criteria

1. Donor should be evaluated for eligibility to donate by an independent physician not directly caring for the patient on study protocol.
2. Donor is willing to sign informed consent allowing the use of the PBSC product for the HSCT of the recipient.
3. Donor cannot be pregnant or lactating and must agree to contraception until after the donation procedure is complete.
4. Testing negative for HIV and viral hepatitis
5. Free of Hb S (defined as Hb S less than 50%) and other hemoglobinopathies that are symptomatic or of clinical significance.
6. Targeted minimum stem cell dose of 5.0 x 10e6 CD34 cells/Kg of recipient weight
7. Fulfills standard criteria for eligibility as a donor for HSCT.

Note: HSCT can be deleterious for the developing fetus and pregnant mother due to the conditioning regimen, GVHD prophylaxis and treatment. Agents used in this study such as cyclophosphamide are pregnancy risk factor category D. Sirolimus is pregnancy risk factor category C. Radiotherapy also used (TBI) is a well-known teratogenic agent. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for at least 1 year post transplant.

Finally, pregnancy and lactation restrictions and contraception requirements are also applicable to the donor. Filgrastim or other G-CSF analogous are pregnancy risk factor category C. The restriction lasts for 4 weeks after stem cell donation.

Exclusion Criteria:

1. Pulmonary dysfunction defined as DLCO (corrected for hemoglobin and alveolar volume) < 40% of predicted OR baseline oxygen saturation of <85% or PaO2 <70.
2. Severe cardiac dysfunction defined as ejection fraction <35%.
3. Impaired renal function defined as GFR <40.
4. Hepatic dysfunction defined as bridging (portal to portal) fibrosis or cirrhosis of the liver OR transaminases >5x ULN for age.
5. Clinical stroke within 6 months of anticipated transplant
6. Karnofsky performance score < 50%
7. HIV infection
8. Uncontrolled viral, bacterial, fungal, or protozoal infection at the time of study enrollment.
9. Have circulating HAMA noted on initial screening.
10. Have received prior radiation to maximally tolerated levels to any critical normal organs
11. Patients with unspecified chronic toxicity serious enough to detrimentally affect the patient's capacity to tolerate HSCT.
12. Patients' unable to understand the nature and risks inherent in the HSCT process.
13. History of non-compliance severe enough in the estimation of the treating team to preclude the patient from undergoing unrelated donor transplantation.
14. Patient is pregnant or lactating.
15. Inability to provide adequate transfusion support or increased risk immunohematological complications due presence of anti-RBC antibody against stem cell donor.
16. Patients with any history of radiation therapy.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2030-03-12 (Estimated); Study Completion 2032-03-12 (Estimated)

PRIMARY OUTCOMES:
Graft failure rate | 42 days after blood stem cell (PB) transplantation
  Graft failure defined as having had a primary or secondary graft failure by 42 days after blood stem cell (PB) transplantation. Primary graft failure is defined as failure to achieve an absolute neutrophil count (ANC) of >500/ μL by 42 days after blood stem cell (PB) transplantation or a total donor chimerism of >5%. Secondary graft failure is defined as cytopenias after initial engraftment (ANC <500/μL) and a total donor cell chimerism decreasing to less than 5%.

SECONDARY OUTCOMES:
Event-free survival (EFS) Rate | Duration of study, up to 7 years
  Event-free survival is defined as the time from treatment initiation to the occurrence of primary graft failure, death, Graft-versus-Host Disease (GVHD) Grade III-IV, whichever comes first. Patients without events will be censored at the time of last follow-up assessment.
Time to engraftment of Neutrophils | Up to 7 years
  Time to neutrophil engraftment is defined as the first of 3 measurements on consecutive days when the patient has an absolute neutrophil count of 500/μL after conditioning.
Time to engraftment of Platelets | Up to 7 years
  Time to platelet engraftment will be defined as the first day of a minimum of 3 measurements on different days that the patient has achieved a platelet count > 50,000/μL AND did not receive a platelet transfusion in the previous 7 days. The exception is the case in which a subject is given a platelet transfusion specifically to achieve a platelet threshold to allow an elective invasive procedure, such as a central catheter removal. Time from treatment initiation to successful donor cell engraftment defined as having achieved > 50% total PMC donor cell chimerism upon successful engraftment at day +30 or upon meeting ANC and Plt engraftment whatever occurs first.
Incidence of Graft-versus-Host Disease (GVHD) of any grade | Up to 7 years
  Incidence of acute and chronic GVHD of any grade as evaluated according to the CIBMTR and NIH criteria respectively.
Incidence of other transplant related toxicities | 12 Months Post Stem Cell Transplant
  Incidence of other transplant related toxicities, including Veno-occlusive disease (VOD), Idiopathic pneumonia syndrome (IPS), Central nervous system (CNS) toxicity, or Posterior reversible encephalopathy syndrome (PRES).
Incidence of significant transplant-related infections | 12 Months Post Stem Cell Transplant
  Significant infections will be recorded including but not limited to bacterial or fungal sepsis, CMV reactivation with/without clinical disease, adenovirus infection, EBV reactivation with or without PTLD, other significant viral reactivations or community-acquired viral infections and invasive mold infections.
Number of participants with donor chimerism >5% | 100 days post-transplant and 1 year post transplant by STR
  Chimerism is a measure of the engraftment of donor cells within the recipient and is expressed as the percentage ratio between the number of donor cells and recipient cells. Chimerism will be determined by Short Tandem Repeat analysis.
Percentage of Participants who Achieve Immune Reconstitution | 12 Months Post Stem Cell Transplant
  Peripheral blood quantitative assessment of CD3+, CD4+, CD8+, CD19+, and CD16+/56+ lymphocytes will be assessed by flow cytometry. In addition, quantitative immunoglobulins will be measured for IgA, IgM and IgG. These will be performed at Day +60 (±10 days) as well as at 1 year (+/- 2 weeks) and after long term follow up at the discretion of the investigator. Descriptive statistics will be used to describe the percentage of patients who are able to achieve reconstitution of important lymphocyte subsets and B cell function at the defined timepoint above.
Follicle-stimulating hormone (FSH) titer | At study inclusion and at 1 year post-transplant
  To assess the impact of the conditioning on fertility, FSH titers will be measured.
Luteinizing hormone (LH) titer | At study inclusion and at 1 year post-transplant
  To assess the impact of the conditioning on fertility, LH titers will be measured.
Anti-Müllerian Hormone (AMH) titer | At study inclusion and at 1 year post-transplant
  To assess the impact of the conditioning on fertility, AMH titers will be measured
Testosterone titer | At study inclusion and at 1 year post-transplant
  To assess the impact of the conditioning on fertility, testosterone titers will be measured.
Sperm titer | At study inclusion and at 1 year post-transplant
  To assess the impact of the conditioning on fertility, sperm titers will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Y Mapara, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided